CLINICAL TRIAL: NCT01296464
Title: Duration of Motor Response After Administration of Experimental Levodopa/Carbidopa/Entacapone Treatment Regimens Compared to Standard Treatment (Stalevo®);a Randomised,Double-blind,Crossover,Multicentre,Single Dose Study in Patients With Parkinson?s Disease and Wearing-off Symptoms
Brief Title: Comparing Different Levodopa/Carbidopa/Entacapone Treatment Regimens
Acronym: PARTEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2939136
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Motor response; Wearing-off
MeSH Terms: conditions — Parkinson Disease | interventions — Carbidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stalevo (Experimental): levodopa/carbidopa/entacapone
  Interventions: Drug: Carbidopa
- Placebo (Placebo Comparator)
  Interventions: Drug: Carbidopa

INTERVENTIONS:
Drug: Carbidopa — Capsules

SUMMARY:
The primary objective is to assess the effect of a single dose of two experimental levodopa/carbidopa/entacapone (L/C/E) treatment regimens versus standard L/C/E treatment regimen in Parkinson's disease (PD) patients with end-of-dose motor fluctuations in terms of duration of motor response after the first morning dose of levodopa. The secondary objective is to evaluate the safety of the L/C/E treatment regimens in patients with PD.

DETAILED DESCRIPTION:
This is a randomised, double-blind, 3-period crossover study comparing the effects of a single dose of two L/C/E treatment regimens (A and B) and standard L/C/E treatment regimen (Stalevo) on the duration of motor response in PD patients with wearing-off symptoms after the first morning dose of levodopa.

The study consists of a screening visit, 3 treatment visits and an end-of-study visit. Within 14 days of the screening visit, the patients will receive a single morning dose of study drug (either of the two L/C/E treatment regimens) or Stalevo. The order of the 3 treatment periods will be randomised according to a crossover design and the duration of each period is 2 days, followed by a wash-out period (1-9 days) during which the patients will be on their individual standard PD treatment.

Before each study day, patients will arrive at the study centre in the previous evening. The patients' own standard PD treatments will be discontinued at the latest by 22:00 to be continued after completion of the motor part (part III) of the Unified Parkinson's Disease Rating Scale (UPDRS III) next day. After completion of the UPDRS III, patients will return to their own standard PD treatments. Duration of the study will be 2 to 7 weeks per patient, depending on the length of the screening and wash-out periods.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* Male or female patients with idiopathic PD according to the United Kingdom brain bank criteria with end-of-dose motor fluctuations
* Hoehn and Yahr stage 2-4 performed during the "ON" state.
* Duration of response between 1.5 and 4 hours (based on medical history) to the patient's first morning dose of levodopa/dopa decarboxylase inhibitor (DDCI) with or without entacapone.
* Treatment with 3-8 daily doses of levodopa/DDCI with or without entacapone with a total daily levodopa dose in the range of 300-1200 mg. One evening dose of controlled-release formulation of levodopa/DDCI is allowed provided that it is included in the total of 3-8 daily doses of levodopa/DDCI mentioned above.
* Unchanged levodopa/DDCI with or without entacapone and other antiparkinsonian medication(dopamine agonists, monoamine oxidase [MAO] B inhibitor, amantadine and/or anticholinergics with approved doses), if any, for at least 6 weeks prior to the screening visit.
* Age of 30 years or above

Exclusion Criteria:

* Secondary or atypical parkinsonism.
* Use of tolcapone within 6 weeks prior to the first treatment period.
* Previous tolerability problems with entacapone or tolcapone.
* Concomitant treatment with apomorphine, MAO-A inhibitors or nonselective MAO inhibitors.
* Concomitant treatment with drugs having antidopaminergic action including alpha-methyldopa, reserpine and antipsychotic drugs (also D2 receptor blocking antiemetics except domperidone). As an exception, an evening dose of an atypical antipsychotic is allowed.
* Use of any iron preparations.
* Intensity of dyskinesias which would, in the opinion of the investigator, interfere with the interpretation of motor part (part III of the Unified Parkinson's Disease Rating Scale (UPDRS III) scoring during the levodopa challenge test.
* Currently active hallucinations.
* Severe orthostatic hypotension as judged by the investigator.
* Mini-Mental State Examination (MMSE) score < 26
* History of neuroleptic malignant syndrome (NMS) and/or non-traumatic rhabdomyolysis.
* Past or current treatment with deep brain stimulation (DBS) or other surgical treatment for PD.
* Treatment with levodopa or dopamine agonist infusion or injection
* Active malignancy, narrow-angle glaucoma or pheochromocytoma.
* Clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, neurological or psychiatric disorder or any other major concurrent illness that in the opinion of the investigator would interfere with the interpretation of the study results or constitute a health risk for the subject if he/she takes part into the study.
* Alanine aminotransferase or aspartate aminotransferase > upper limit of normal at screening.
* Any other abnormal value of laboratory, vital signs or electrocardiogra (ECG) which would in the opinion of the investigator interfere with the interpretation of the study results or cause health risk for the subject if he/she takes part into the study.
* Female patients of childbearing potential (i.e. menstruating or less than 2 years postmenopausal) if they are not using proper contraception (hormonal contraception, intrauterine device [IUD] or surgical sterilisation, spermicidal foam in conjunction with condom on male partner).
* Patients with pre-planned elective surgery.
* Known hypersensitivity to active substances or to any of the excipients of the study drugs.
* Participation in a drug study within 60 days prior to entry to this study.
* Any other condition that in the opinion of the investigator would interfere with the interpretation of the study results or constitute a health risk for the subject if he/she takes part into the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Duration of motor response by UPDRS III | 20 minute intervals
  Statistical method for the primary comparison will be analysis of variance (ANOVA) with the following grouping factors: treatment, sequence, subject, and period. Differences between Stalevo and treatment regimen A will be evaluated using orthogonal contrasts with 5% significance level.

CONTACTS AND LOCATIONS:
Overall Officials: Vilho Myllylä, Prof, Principal Investigator — Oulu Deaconess Instutute
Locations (5):
- Finland (3):
  - Kanta-Hämeen keskussairaala, Hämeenlinna
  - ODL Terveys Oy (ODL), Oulu
  - Porin Lääkäritalo, Pori
- Sweden (2):
  - Länssjukhuset Ryhov, Medicin/Neurologmottagningen, Jönköping
  - Karolinska Universitetssjukhuset Solna, Neurologkliniken, Stockholm